CLINICAL TRIAL: NCT03529084
Title: A Randomized, Open-label, Phase III Study of Single Agent Nazartinib Versus Investigator's Choice (Erlotinib or Gefitinib) as First-Line Treatment in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Harboring EGFR Activating Mutations
Brief Title: Phase III Study of Nazartinib (EGF816) Versus Erlotinib/Gefitinib in First-line Locally Advanced / Metastatic NSCLC With EGFR Activating Mutations
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision by Sponsor not to continue with the trial.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEGF816A2302; 2017-003998-34 (EudraCT Number)
Record Dates: First submitted 2018-04-18; First posted 2018-05-18 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Non-small Cell Lung
Keywords: Non small cell lung cancer; NSCLC; EGFR mutation; EGF816; nazartinib; erlotinib; gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nazartinib; Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinded independent review committee for primary endpoint of PFS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EGF816 (Experimental): Investigational treatment arm of EGF816 (nazartinib).
  Interventions: Drug: EFG816
- Investigator's Choice (Active Comparator): Investigator's Choice (erlotinib or gefitinib).
  Interventions: Drug: erlotinib or gefitinib

INTERVENTIONS:
Drug: EFG816 — It will be administered orally daily.
  Other Names: nazartinib
  Arms: EGF816
Drug: erlotinib or gefitinib — Investigator's choice between erlotinib or gefitinib. These will be locally sourced.
  Erlotinib will be administered orally daily. Gefitinib will be administered orally daily.
  Arms: Investigator's Choice

SUMMARY:
This is a phase III, open label, randomized controlled multi-center global study designed to evaluate the safety and efficacy of single agent nazartinib (EGF816) compared with investigator's choice (erlotinib or gefitinib) in patients with locally advanced or metastatic NSCLC who are treatment naïve and whose tumors harbor EGFR activating mutations (L858R or ex19del).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any screening procedures.
* Histologically documented locally advanced or metastatic, stage IIIB/ IIIC or stage IV NSCLC with documented EGFR activating mutation (L858R or ex19del)
* Provision of a tumor tissue sample to allow for retrospective analysis of EGFR mutation status
* No prior treatment with any systemic antineoplastic therapy in the advanced setting
* Recovered from all toxicities related to prior treatment
* Presence of at least one measurable lesion according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance ≤1
* Meet the following laboratory values at the screening visit:

  * Absolute Neutrophil Count ≥1.5 x 109/L
  * Platelets ≥75 x 109/L
  * Hemoglobin (Hgb) ≥9 g/dL
  * Creatinine Clearance ≥ 45 mL/min using Cockcroft-Gault formula
  * Total bilirubin ≤1.5 x ULN
  * Aspartate transaminase (AST) ≤ 3.0 x ULN, except for patients with liver metastasis, who may only be included if AST ≤5.0 x ULN
  * Alanine transaminase (ALT) ≤ 3.0 x ULN, except for patients with liver metastasis, who may only be included if ALT ≤5.0 x ULN

Exclusion Criteria:

* Prior treatment with EGFR-TKI.
* Known T790M positive mutation. Any other known EGFR activating mutations other than L858R or ex19del. Patients whose tumors harbor other EGFR mutations concurrent with L858R or ex19del EGFR mutations are eligible.
* Symptomatic brain metastases
* History of interstitial lung disease or interstitial pneumonitis
* Any medical condition that would, in the investigator's judgment, the patient's in the study due to safety concerns, compliance with clinical study procedures or interpretation of study results
* Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years..
* Presence of clinically significant ophthalmologic abnormalities
* Bullous and exfoliative skin disorders of any grade
* Presence or history of microangiopathic hemolytic anemia with thrombocytopenia.
* Known history of testing positive for human immunodeficiency virus (HIV) infection
* Cardiac or cardiac repolarization abnormality
* Major surgery: ≤4 weeks to starting study treatment or who have not recovered from side effects of such procedure.
* Unable or unwilling to swallow tablets or capsules
* Female patients who are either pregnant or nursing
* Women of child bearing potential who refuse or are not able to use a highly effective method of contraception as defined in the study protocol.
* Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of study treatment.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-24 (Estimated); Primary Completion 2020-08-13 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by Blinded independent review committee (BIRC) | Approximately 3 years
  PFS using central BIRC assessment according to RECIST 1.1, is defined as the time from the date of randomization to the date of the first documented progression (as assessed by BIRC per RECIST 1.1) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | Approximately 6 years
  Overall survival is defined as the time from date of randomization to date of death due to any cause.
PFS by investigator | Approximately 3 years
  PFS by Investigator assessment according to RECIST 1.1, is defined as the time from the date of randomization to the date of the first documented progression (as assessed by Investigator per RECIST 1.1) or death due to any cause, whichever occurs first.
PFS after next-line of treatment (PFS2) using investigator assessment according to RECIST 1.1 | Approximately 4 years
  PFS after next-line of treatment (PFS2) using investigator assessment according to RECIST 1.1 is defined as time from date of randomization to the first documented disease progression (clinical or radiologic) as per investigator assessment on next-line therapy or death from any cause, whichever occurs first.
Time to progression in Central Nervous System (CNS) per central neuro-radiologist BIRC | Approximately 3 years
  Time to progression in CNS, defined as time from date of randomization to the date of first documented progression of brain metastases as assessed by central neuro-radiologist BIRC per modified RECIST 1.1 for patients with at least one non-measurable and/or measurable lesion in the brain at baseline.
Overall response rate (ORR) by central BIRC | Approximately 3 years
  ORR in accordance with RECIST 1.1. ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR)
Duration of response (DOR) by central BIRC | Approximately 3 years
  DOR is defined as the time from date of first documented response (CR and PR) to the date of the first documented progression or death due to underlying cancer, whichever occurs first.
Disease control rate (DCR) by central BIRC | Approximately 3 years
  DCR is defined as the percentage of participants with BOR of CR, PR, or stable disease (SD).
Time to response (TTR) by central BIRC | Approximately 3 years
  TTR is defined as the time from the date of randomization to the first documented response CR or PR.
CNS ORR per central neuro-radiologist BIRC | Approximately 3 years
  CNS ORR in patients with brain metastases who have measurable disease in the brain at baseline review per modified RECIST 1.1
CNS DoR per central neuro-radiologist BIRC | Approximately 3 years
  CNS DoR in patients with brain metastases who have measurable disease in the brain at baseline per modified RECIST 1.1
Charactise Plasma PK (Cmax) of EGF816 | Day 1 of Cycles 1 to 6 inclusive (21 day cycle)
  Peak plasma concentration (Cmax) of EGF816 and its metabolite (LMI258)
Charactise Plasma PK (AUC) of EGF816 | Day 1 of Cycles 1 to 6 inclusive (21 day cycle)
  Area under the plasma concentration versus time curve (AUC) of EGF816 and its metabolite (LMI258)
Charactise Plasma PK (t1/2) of EGF816 | Day 1 of Cycles 1 to 6 inclusive (21 day cycle)
  Elimination half life (t1/2) of EGF816 and its metabolite (LMI258)
Patient Reported Outcome: Health Related Quality of Life (HRQoL) as measured by QLQ-C30 Questionnaire | Approximately 4 years
  HRQoL as measured by European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 quality of life score
Patient Reported Outcome: Health Related Quality of Life (HRQoL) as measured by QLQ-LC13 Questionnaire | Approximately 4 years
  HRQoL as measured by European Organization for Research and Treatment of Cancer (EORTC) QLQ-LC13 quality of life score
Patient Reported Outcome: Health Related Quality of Life (HRQoL) as measured by EuroQoL-5 Dimension-5 (EQ-5D-5L) Questionnaire | Approximately 4 years
  Global health status/quality of life score of the EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.